CLINICAL TRIAL: NCT03845049
Title: Comparative Multicenter Randomized Study of Aflibercept Versus Placebo in Macular Telangiectasia Type 1
Acronym: TELeMAC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: very rare disease, many difficulties in recruiting patients, inclusion rate far too slow, making it impossible to meet the main objective within a reasonable timeframe. the sponsor therefore decided to stop the study.
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CREUZOT PHRC N 2017
Record Dates: First submitted 2019-02-15; First posted 2019-02-19 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Macular Telangiectasia
MeSH Terms: interventions — aflibercept; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group aflibercept (Experimental)
  Interventions: Other: Inclusion examinations; Drug: Aflibercept Injection [Eylea]; Other: Examinations during study (every month)
- control group (Placebo Comparator)
  Interventions: Other: Inclusion examinations; Drug: SHAM injection; Other: Examinations during study (every month)

INTERVENTIONS:
Other: Inclusion examinations — Pregnancy test, Visual acuity, ocular pressure, color retinophotography, OCT-SD (the Heidelberg SDOCT Spectralis, or the Cirrus HD-OCT, model 5000, Zeiss), OCT-angiography and fluorescein angiography and wide-field angiogram
Drug: Aflibercept Injection [Eylea] — Intravitreal injection of aflibercept at inclusion, M1, M2, M3 and M4. An additional injection may be planned for M5, on the decision of the clinician and on clinical arguments only.
  Arms: group aflibercept
Drug: SHAM injection — Intravitreal injection of SHAM at inclusion, M1, M2, M3 and M4. An additional injection may be planned for M5, on the decision of the clinician and on clinical arguments only.
  Arms: control group
Other: Examinations during study (every month) — visual acuity, ocular pressure, OCT-SD, OCT-angiography and ocular fundus and a pregnancy test at M6

SUMMARY:
Idiopathic juxtafoveal telangiectasia type 1 is a rare unilateral disease that mostly affects men before 50 years of age. Mac Tel 1 are characterized by microvascular telangiectasia and increased tortuosity of the macular capillary network on the temporal part of the fovea that can be identified on fundus examination. It can be associated with peripheral vascular changes, similar to manifestations of Coats' disease. It can be complicated by macular edema due to leakage from microvascular ectasia. When associated with visual loss, macular edema can be treated with different strategies although there is no consensus about the best approach. Laser can be performed on leaky aneurysms with questionable long term efficacy and potential irreversible adverse effects. Recently, anti-VEGF agents have been put forward as particularly good candidates to treat this macular edema, as observed in vein occlusion or diabetic macular edema. Indeed, in limited case series, the first anti-VEGF agents (ranibizumab and bevacizumab) showed mitigated results. More recently, authors have reported some favorable results with aflibercept in patients refractory to other anti-VEGF agents. Indeed a recent study reported both good anatomical and functional results in macular edema due to Mac Tel 1 in a non-comparative study that included 8 patients and carried out a concomitant quantification of growth factors. As an explanation, the authors found that levels of placental growth factor (PlGF), which is targeted by aflibercept but not by other anti-VEGF agents, were decreased after treatment. Moreover, PlGF correlated with capillary plexus densities assessed by OCTA. The aim of this study is thus to assess the efficacy of a 6 months treatment by aflibercept compared to placebo in macular edema linked to Mac Tel 1 with a multicenter double-blind randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient who have given their written informed consent
* Patient major
* Patient with idiopathic macular telangiectasia type 1 identified at least 4 months previously, with or without peripheral exudative abnormalities
* Patient with macular edema more than 320 μm confirmed by a blind review of SD-OCT images
* Patient with best-corrected ETDRS visual acuity between strictly24 and 79 letters
* Patient meeting at least 1 of the following criteria:
* Patient naive to any treatment
* Patient with a contraindication for laser photocoagulation
* Patient with persistence of macular edema after treatment with anti-VEGF (including aflibercept) administered more than 4 months previously
* Patient with persistence of macular edema after laser photocoagulation treatment more than 4 months previously
* Patient with persistence of macular edema after treatment with corticosteroids administered more than 6 months previously
* Patient with an assessment by the treating ophthalmologist that focal coagulation (for both groups) and anti-VEGF treatment (for the placebo group) could be safely deferred for 6 months
* Woman of childbearing potential (WOCBP)* must commit to consider and use an efficient method of birth control during the trial and at least 3 months after the last aflibercept/SHAM administration

Exclusion Criteria:

* Patient not affiliated to a national health insurance scheme
* Patient subject to a measure of legal protection (guardianship, tutorship)
* Patient subject to a court order
* Patient pregnant, parturient or nursing women (WOCBP)*
* Patient incapable of expressing consent
* Patient with edema linked to conditions other than macular telangiectasia (namely retinal vein occlusion, diabetic retinopathy, ocular ischemic syndrome, sickle-cell anemia, maculopathy, hypertensive retinopathy…)
* Patient presenting any cardiovascular eventwithin 6 months before inclusion
* Poor media clarity, which can prevent adequate fundus imaging
* Patient with hypersensitivity to the active substance (aflibercept) or to any of the excipients of EYLEA®
* Patient with active or suspected ocular or periocular infection or severe active intraocular inflammation.
* Any history of allergy to the antiseptic used during preparation of the eye for the IVT injection in the investigational site (e.g. povidone iodine or chlorhexidine).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Change in central retinal thickness (CRT) | Between M0 and M6

CONTACTS AND LOCATIONS:
Locations (1):
- CHU dijon Bourgogne, Dijon, France